CLINICAL TRIAL: NCT05000905
Title: A Pilot Study of Assessing and Improving Cognition and Real-World Behavior in Pediatric Cancer Survivors
Brief Title: Improving Cognition and Behavior in Pediatric Cancer Survivors Using a Novel Mindful Attention Training
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 210822; NCI-2022-07364 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-08-09; First posted 2021-08-11 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Cancer
Keywords: Pediatric Cancer Survivor; Attention; Cognitive Control
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Forty participants will be randomized to the Engage intervention (30-session) or low-dose (2-session). Individuals in each active arm will be matched on age and gender.
  An additional thirty participants will be enrolled separately (not randomized) into the no-contact group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adaptive Attention Training (Experimental): Participants will complete approximately 15 hours of an at-home training on a novel adaptive attention training program ('Engage'), which will consist of completing thirty, 30-minute sessions over a total of 6-8 weeks.
  Interventions: Behavioral: Adaptive Attention Training; Behavioral: Questionnaires
- Low-dose Adaptive Attention Training (Active Comparator): Participants will complete approximately 1 hour of at-home training on 'Engage' which consists of two, 30-minute sessions at the beginning and middle of a 6-8 week period.
  Interventions: Behavioral: Adaptive Attention Training; Behavioral: Questionnaires
- No Contact Group (Not Randomized) (Other): An additional thirty participants will be enrolled separately (not randomized) into the no-contact group. Participants in the no-contact group will not complete any study activities for 6-8 weeks after completing the baseline assessments. After this period, participants will be prompted to log into Nexus to complete end of study assessments (same set of assessments administered/completed at baseline).
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Adaptive Attention Training — The training is comprised of a time-based titration of rich audiovisual and sparse audio interactive environments. Training progressively transitions the participants from an immersive and rapid reward setting to a less immersive, sensory impoverished, and slower reward setting. Further, the participants' actions require delayed gratification decisions to accomplish play in the sparse setting, building fronto-parietal control through sustained attention and suppression of ventral-striatal reward impulses.
  Arms: Adaptive Attention Training; Low-dose Adaptive Attention Training
Behavioral: Questionnaires — Computer based assessments measuring attention, memory, daily habits, and mental health

SUMMARY:
This pilot study will evaluate the cognitive and behavioral outcomes of using a novel, adaptive attention training in pediatric cancer survivors.

DETAILED DESCRIPTION:
Pediatric cancer survivors (PCS) often experience attentional difficulties that have downstream effects on their quality of life, academic achievement, and future occupational attainment. As such, the primary goal of this project is to examine the outcomes of a novel, mindful attention training in this population and assess the feasibility of recruitment, retention, and adherence. Specifically, PCS will be randomly assigned to one of two adaptive attention training groups ('Engage') and complete tasks on the device for up to 8 weeks. Participants will also complete pre- and post-training assessments of cognition and behavior.

An additional cohort of no-contact participants will be asked to complete the assessments at baseline and end of study only to assess the feasibility and reliability of the assessment measures. This cohort will be enrolled separately and not randomized.

The investigators hypothesize that completion of 'Engage' training for the randomized cohorts will result in enhanced attentional control beyond the active comparator group that extends to other aspects of cognition in PCS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7-17 at the time of enrollment.
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Ability of individual and legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
4. Normal or corrected-normal vision and hearing.
5. English language fluency (minor participant and parent/guardian).
6. Received radiation therapy to the brain or neck between age 7-17.
7. Patients not on current cancer-related treatment (except supportive care) or those on other current treatments that would not hinder study participation. Patients currently on cancer-related treatments will be discussed with the study team (co-PI Mueller).

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.
2. Motor/perceptual difficulties that prevent computer or tablet use.
3. Current cancer-related treatments that would impact the ability to participate in the study (e.g., current inpatient chemotherapy or intrathecal chemotherapy). Patients on other current treatments will be discussed with the study team (co-PI, Dr. Mueller)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who complete study | Up to 8 weeks
  The proportion of participants who completed the study procedures will be reported by study cohort.

SECONDARY OUTCOMES:
Change in mean performance on a Continuous Performance Task (CPT) over time | Up to 8 weeks
  The CPT is a 23-minute task, where participants are instructed to respond to target stimuli (squares at the top of the screen) and withhold responses to non-target stimuli (squares at the bottom of the screen). Performance will be quantified as: (1) mean reaction times, (2) standard deviation of reaction times (RTV), and (3) d-prime (comparing correct target detections or 'hits' to incorrect non-target detections or 'false alarms').

OTHER OUTCOMES:
Change in sub-test scores on the Adaptive Cognitive Evaluation (ACE) neuropsychological battery | Up to 8 weeks
  The ACE is a mobile cognitive assessment tool, which includes a battery of cognitive control tests for rapid tests of cognition. The sub-tests (or 'modules') in ACE are adapted from standardized tasks to rapidly assess various aspects of cognition, including attention, memory, and multitasking.
Change in mean performance on a computerized Math Fluency Test | Up to 8 weeks
  To assess math fluency, participants solve simple math problems (e.g., addition, subtraction, multiplication) over a 3-minute period. Performance is measured as the number of correct responses.
Change in mean performance on a computerized Reading Fluency Test | Up to 8 weeks
  To assess reading fluency, participants indicate whether sentences are 'True' or 'False' over a 3-minute period. Performance is measured as the number of correct responses.
Change in mean scores on the Mindful Attention Awareness Scale (MAAS) over time | Up to 8 weeks
  The MAAS is a 15-item scale designed to assess a core characteristic of mindfulness by asking participants to respond to statements about everyday experiences on a scale from 1="Almost always" to 6="Almost never". The total score is obtained by averaging the scores of the 15 items, to generate a total score for from 1-6. Greater scores are indicative of a greater level of mindfulness.
Change in mean scores on the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) over time | Up to 8 weeks
  The 14-item scale WEMWBS addresses mental well-being by asking participants to respond to individual items on a scale from 1="None of the time" to 5="All of the time". The total score is obtained by summing the scores for each of the 14 items, to generate a total score ranging from 14-70. Lower scores are indicative of a lower overall well-being.
Change in mean scores on a modified Insomnia Severity Index (ISI) Scale over time | Up to 8 weeks
  The modified ISI consists of the first three of seven items in the full ISI scale. These three questions ask participants about the the severity of their insomnia symptoms on a scale from 0="None" to 4="Very". The total score is obtained by summing the scores for each of the three items, to generate a total score from 0-12. Higher scores are indicative of more insomnia problems.
Change in mean scores on the Child Self-Control Rating Scale (parent rating) over time | Up to 8 weeks
  The Child Self-Control Rating Scale consists of 33 items that assess children's self control. Parents respond to individual items on a 7-point scale. The total score is obtained by summing the scores for each of the 33 items, with a higher score reflecting greater lack of child self-control.
Change in mean performance on a Delay Discounting Task over time | Up to 8 weeks
  The Delay Discounting task is an untimed task, where participants choose between smaller, more immediate rewards and larger, more delayed rewards. Performance will be quantified by comparing choices between smaller/immediate rewards and larger/delayed rewards as the rate of delay discounting (the hyperbolic discounting index).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Anguera, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No